CLINICAL TRIAL: NCT01874067
Title: C-GLOVES: an Evaluation of the Effectiveness of Compression Gloves in Arthritis: a Feasibility Study
Brief Title: C-GLOVES: the Effectiveness of Compression Gloves in Arthritis
Acronym: C-GLOVES
Status: Completed | Type: Observational
Sponsor: University of Salford (Other)
Responsible Party: Principal Investigator, Alison Hammond, Professor in Rheumatology Rehabilitation, University of Salford
Other Study IDs: C-GLOVES v2 26.7.13; 13/EM/0253 (Other: NHS Research Ethics Committee (UK))
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Inflammatory Arthritis; Rheumatoid Arthritis; Hand Osteoarthritis
MeSH Terms: conditions — Arthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Arthritis glove: Early inflammatory, rheumatoid or hand osteoarthritis with hand/wrist swelling and pain
  Interventions: Device: Arthritis glove

INTERVENTIONS:
Device: Arthritis glove — Isotoner three-quarter finger arthritis glove

SUMMARY:
This is a collaborative study with 11 Occupational Therapy (OT) departments in North-West England. The OTs provide arthritis gloves to 25% of out-patients with inflammatory, rheumatoid and osteoarthritis. The pressure applied by the glove(s) may help relieve hand pain, swelling and stiffness. People find they help but there is little research testing this. Of the five small studies published: two found little or no benefit; one found similar effects from arthritis and ordinary thermal gloves; two found some benefits. Testing if gloves work helps therapists and patients judge if they will help.

This is a feasibility study to help us plan a future trial testing if arthritis gloves work for people with arthritis. We aim to find out: the rate we can recruit people to the study; if OTs can assess people's hands and provide gloves as agreed; how many people do we need to take part in a trial; what do people think (if any) is the gloves' most important effect and how long should we test them for? We will analyse the data to see what effect the gloves have.

The study will last 12 months. People will get arthritis gloves as part of their usual care. The OTs have agreed a standard way of assessing and providing the gloves to ensure best practice across departments. The assessments include: difficulties using hands, pain and stiffness levels, and measuring hand and finger joint size and movement. People can take part if they: have one of the three types of arthritis; are willing to wear Isotoner three-quarter length gloves; can attend the usual 4 week review appointment for re-assessment; will allow us to use their anonymized hand assessments. We will also interview some people about their views of the assessment and their treatment. Each patient will be involved for 4-8 weeks.

DETAILED DESCRIPTION:
Design:

An observational study of usual care providing arthritis gloves with pre- and 4 weeks post-treatment assessment. Participants are screened and recruited (if eligible and consenting) as they attend for glove provision as part of routine care. (Participants are not randomly assigned).

Intervention:

Three-quarter length finger Isotoner glove(s) for one or both hands, as required. The participating OTs determine if patients meet their agreed criteria for gloves as part of usual care. Usually at the same appointment the OT then assesses for and provides these using the assessment and treatment protocols agreed by North West England College of Occupational Therapists Specialist Section - Rheumatology (NWCOTSS-R) members as part of their usual care. Four weeks later, patients attend a review appointment (as part of their usual care) for re-assessment of their hand(s), and to identify any effects the gloves have had and if any problems arose meaning glove wear should be stopped or the wear regimen altered. Normally the patient attends for two appointments only.

Occupational therapist (OT) training

The members of the NWCOTSS-R group agreed the glove provision criteria, hand assessment and treatment protocols and glove instruction sheet in order to improve standards of usual care in glove provision across Rheumatology OT departments. Prior to recruitment commencing, the participating OTs attended a training meeting to ensure they:

* performed the hand assessments (i.e. swelling, finger flexion and Grip Ability Test) reliably.
* Know how to correctly size and fit the gloves following training by an experienced Rheumatology OT
* understand the study procedures, know how to take study specific consent and complete study site documentation.

A standardised assessment kit and manual was provided to the OTs by the University research centre.

Study criteria:

Inclusion:

1. Meet the criteria agreed by NWCOTSS-R members for receiving compression gloves as part of usual OT care.
2. Adults with either:

i. early inflammatory, probable or definite RA, diagnosed by a Rheumatology Consultant ii. hand OA, diagnosed by a GP, Consultant or Advanced Practitioner.

c) Willing and able to wear three-quarter length Isotoner glove(s), following the glove fitting process.

d) Willing to attend for the glove review appointment (part of usual care) approximately four weeks following glove provision.

Exclusion:

e) Has a terminal illness, or other health or personal issues, such that the OT considers the patient's participation may be an undue burden.

f) Has any other condition which could alter hand symptoms and function between assessments (eg stroke, multiple sclerosis)

g) In early IA/RA or hand OA: received an intra-articular or intra-muscular steroid injection or started a new anti-inflammatory drug within the last 4 weeks

h) In established RA only: started a new DMARD within the last 6 weeks

Sample size:

40 people from each of the: early IA or RA; and Hand OA, condition groups will be recruited. As this is a feasibility study no sample size has been calculated.

ELIGIBILITY:
Inclusion Criteria:

* experiencing hand pain and swelling

Exclusion Criteria:

* unable to give informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatology Occupational Therapy and Hand Therapy out-patient departments
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Hand pain on movement | 4 weeks
  10 point numeric rating scale of hand pain during moderate activities (eg housework, gardening, work) with end points of no to severe pain

SECONDARY OUTCOMES:
Measure of Activity Performance in the Hand: patient reported outcome | 4 weeks
  patient reported outcome of hand function
Grip Ability Test | 4 weeks
  objective measure of hand function

CONTACTS AND LOCATIONS:
Overall Officials: Alison Hammond, PhD, Principal Investigator — University of Salford
Locations (5):
- United Kingdom (5):
  - Occupational Therapy, Leighton Hospital, Crewe, Cheshire
  - Occupational Therapy, Victoria Infirmary, Northwich, Cheshire
  - Occupational Therapy Department, Stepping Hill Hospital, Stockport, Greater Manchester
  - Ocupational Therapy, St Helens Hospital, St Helens, Knowsley
  - Occupational Therapy, Southport District General Hospital, Southport, Merseyside

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hammond A, Prior Y, Jones V, Dooley M, Hough Y, Jacklin A. A Pre-Test Post-test pilot trial of compression gloves in early inflammatory and rheumatoid arthritis. Rheumatology 54(S1):i111-112, 2015. doi:10.1093/rheumatology/kev089.045
- [Background] Hammond A, Prior Y, Jones V, Dooley M, Hough Y, Jacklin A. The Effect of Compression Gloves in Hand Osteoarthritis: A Pre-Pest-Test Trial. Arthritis and Rheumatism 66(11 Supplement): S436, 2014
- [Background] Hammond A, Prior Y. Compression gloves for patients with hand arthritis (C-GLOVES): A feasibility study. Hand Ther. 2021 Mar;26(1):26-37. doi: 10.1177/1758998320986829. Epub 2021 Jan 12. PMID 37905193
- [Background] Hammond A, Prior Y. Arthritis glove provision in rheumatoid arthritis and hand osteoarthritis: A survey of United Kingdom rheumatology occupational therapists. Hand Ther. 2022 Mar;27(1):3-13. doi: 10.1177/17589983211060620. Epub 2022 Jan 5. PMID 37904793